CLINICAL TRIAL: NCT02186184
Title: Effect of Orthokeratology on Myopia Progression in Chinese Children
Brief Title: Effect of Orthokeratology Versus Spectacles on Myopia Progression in Chinese Children: A Crossover Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Shi-Ming Li, Dr., Beijing Tongren Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CB504601
Record Dates: First submitted 2014-06-29; First posted 2014-07-10 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Myopia
Keywords: Myopia progression; Orthokeratology
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orthokeratology in the first year (Experimental): The participants would wear orthokeratology in the first year and then switch to spectacle in the second year
  Interventions: Device: Orthokeratology; Device: Spectacle
- Spectacle in the first year (Active Comparator): The participants would wear spectacle in the first year and then changed to orthokeratology in the second year
  Interventions: Device: Orthokeratology; Device: Spectacle

INTERVENTIONS:
Device: Orthokeratology
Device: Spectacle
  Other Names: Glasses

SUMMARY:
Orthokeratology is becoming popular for the treatment of myopia children. Many studies have shown that orthokeratology is effective in temporarily reducing refractive error, and is also helpful for controlling myopia progression. However, the mechanism for its slowing myopia progression and rebound effect after the treatment have not been clearly studied. In addition, the effect of orthokeratology among Chinese children has not been evaluated with randomized controlled trial.This study is to assess the effect of orthokeratology versus spectacles on myopia progression in school-aged Chinese children during two years.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 7 Years to 14 Years
* Genders Eligible for Study: Both
* Visual acuity 20/20 or better in each eye
* Spherical error ranging from -0.5 D to -5.0 D and astigmatism less than 1.5 D in each eye, anisometropia less than 1.0 D between the two eyes
* No strabismus, amblyopia and any other ocular or systematic diseases that may affect refractive development

Exclusion Criteria:

* Currently or history using other interventions to control myopia progression (acupuncture, drugs, contact lens, ear needles and so on)
* Unable to cooperate with the ocular examination,questionnaire survey,or orthokeratology wearing

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Refraction | Change from baseline at 1 year
  The participants will be measured for their cycloplegic central refractive error before and after wearing the orthokeratology. Peripheral refraction will also be measured by WAM-5500.
Axial length | Change from baseline at 1 year
  The Lenstar will be used to measure the axial length.
Refraction | Change from baseline at 2 years
Axial length | Change from baseline at 2 years

SECONDARY OUTCOMES:
Tear film break up time(BUT) | Change from baseline at 1 year
Self evaluation of comfortableness | Change from baseline at 1 year
Corneal endothelial cell density | Change from baseline at 1 year
Tear film break up time(BUT) | Change from baseline at 2 years
Self evaluation of comfortness | Change from baseline at 2 years
Corneal endothelial cell density | Change from baseline at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, MD,PhD, Principal Investigator — Beijing Tongren Eye Center, Beijing Tongren Hospital, Capital Medical University
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China